CLINICAL TRIAL: NCT02801552
Title: Regenerative Endodontic Procedure of Immature Permanent Teeth With Apical Periodontitis Using Platelet-rich Fibrin : A Pilot Randomized Controlled Trial
Brief Title: Regenerative Endodontic Procedure of Immature Permanent Teeth With Apical Periodontitis Using PRF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Xiaojing Huang, DDS, PhD, Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JS14031
Record Dates: First submitted 2016-06-12; First posted 2016-06-16 (Estimated); Last update posted 2021-09-05 (Actual); Status verified 2021-09

CONDITIONS: Periapical Periodontitis; Tooth Diseases; Stomatognathic Diseases
Keywords: regenerative endodontic treatment; platelet-rich fibrin; Immature permanent tooth; apical periodontitis
MeSH Terms: conditions — Periapical Periodontitis; Tooth Diseases; Stomatognathic Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Regenerative Endodontic Procedure + PRF (Experimental): Visit 1: root canal dressing with triple antibiotic paste. Visit 2: a 5 ml sample of whole blood was drawn intravenously from the patient's forearm. The blood sample is centrifuged at 400 g for 10 min. The prepared PRF membrane is cut into segments, the fragments are placed into the canal space. The coronal is sealed mineral trioxide aggregate and composite resin.
  Interventions: Device: PRF
- Regenerative Endodontic Procedure (No Intervention): Regenerative Endodontic Procedure Visit 1: root canal dressing with triple antibiotic paste. Visit 2: Blood clot formation is induced in the root canal after disinfection. No PRF was used in this group. Then the canal access is sealed with mineral trioxide aggregate and composite resin.

INTERVENTIONS:
Device: PRF — Regenerative Endodontic Procedure with PRF: autologous PRF will be used instead of blood clot in the second vist.
  Other Names: mineral trioxide aggregate
  Arms: Regenerative Endodontic Procedure + PRF

SUMMARY:
This study evaluates the clinical effect of regenerative endodontic procedure using PRF in immature permanent teeth with apical periodontitis. Half of participants will receive the PRF instead of blood clots in the regenerative endodontic procedure, while the other half will receive a blood clots in the regenerative endodontic procedure.

DETAILED DESCRIPTION:
The conventional method of regenerative endodontic procedure using a blood clot as scaffold materials has shown successful results. However, it is very difficult to induce bleeding and place mineral trioxide aggregate over a blood clot. Platelet-rich fibrin (PRF), a second-generation platelet concentrate. PRF is a matrix of autologous fibrin containing a large quantity of platelets, growth factors and leukocytes. PRF preparation technique is very simple, inexpensive and doesn't require any chemical agents. The purpose of this study is to test the hypothesis that the use of PRF in regenerative endodontic procedure of immature permanent teeth with apical periodontitis will accelerate periapical bone healing and stimulate the root maturation.

ELIGIBILITY:
Inclusion Criteria:

* Between 6 and 18 years of age
* Provision of Informed Consent
* Cooperative in the dental chair
* Permanent immature teeth with apical periodontitis and incomplete root development

Exclusion Criteria:

* Have a medical history that may complicate treatment
* Unlikely to be able to comply with the study procedures

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2019-11 (Actual); Study Completion 2020-02 (Actual)

PRIMARY OUTCOMES:
Evidence of periapical healing | 12 months

SECONDARY OUTCOMES:
Evidence of root development | 24 months
Evidence of pulp sensibility | 24 months
  a positive response to pulp sensibility tests include cold test and electric pulp testing

CONTACTS AND LOCATIONS:
Overall Officials: Xiaojing Huang, PhD, Study Chair — School and Hospital of Stomatology, Fujian Medical University
Locations (1):
- School and Hospital of Stomatology, Fujian Medical University, Fuzhou, Fujian, China

IPD SHARING:
Plan to Share IPD: No